CLINICAL TRIAL: NCT03053986
Title: A Double-blind, Placebo-controlled, Randomized Clinical Trial on the Metabolic and Vascular Effects of a Dietary Supplementation With Apple Polyphenols in Overweight Subjects
Brief Title: Effect of Apple Polyphenols on Vascular Oxidative Stress and Endothelium Function Study (APP trial_2016)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Full Professor of Internal Medicine, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APP trial_2016
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apple polyphenols (Active Comparator): White capsule containing 300 mg of apple extract (Malus Domestica) with glycosilated polyphenols (≥90%) including glycosilated phloritzin (15-30%), chlorogenic acid (10-25%) and quercetin (15-25%)
  Interventions: Dietary Supplement: Apple polyphenols
- Placebo (Placebo Comparator): Indistinguishable capsules with similar dimension, colour, odour and taste
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Apple polyphenols — 1 tablet per day at evening before sleeping
  Arms: Apple polyphenols
Other: Placebo — 1 tablet per day at evening before sleeping
  Arms: Placebo

SUMMARY:
Apple polyphenols are mostly acknowledged for their hypoglycaemic properties, but represent an apple active fraction with many pharmacological functions. The study aim was to examine their effect on uricemia and endothelial function in a sample of overweight subjects. This was a two-phases study. The in vitro experiment aimed to evaluate the apple polyphenols' ability to lower uric acid in comparison with allopurinol. The in vivo study consisted in a randomized, double-blind, parallel placebo-controlled clinical trial involving 62 overweight volunteers with suboptimal values of fasting plasma glucose (100 mg/dL≤FPG≤125 mg/dL), randomized to be treated with 300 mg apple polyphenols or placebo for 8 weeks.

DETAILED DESCRIPTION:
The study included a 2-week run-in period of diet standardization and an 8-week treatment period. At enrolment, patients were given standard behavioural and qualitative dietary suggestions to correct their unhealthy habits. In particular, subjects were strongly recommended to follow the general indications of a Mediterranean diet, avoiding an excessive intake of diary and red meat derived products and reducing the dietary excesses, in order to maintain an overall balanced diet for the entire duration of the study. Individuals were also encouraged to increase their physical activity by walking briskly or cycling from 3 to 5 times for week, at least 20 minutes every time.

The study fully complied with the ethical guidelines of the Declaration of Helsinki. The study protocol was approved by the Ethical Committee of the University of Bologna. All patients signed a written informed consent to participate.

After 2 weeks of diet standardization, the enrolled subjects were allocated to the treatment with an indistinguishable pill of placebo or an active product, containing 300 mg of apple extract (Malus Domestica) with glycosilated polyphenols (≥90%) including glycosilated phloritzin (15-30%), chlorogenic acid (10-25%) and quercetin (15-25%) (kindly provided by Amitalia Srl, Solara, MI, Italy). Patients were asked to take the pills regularly, every day early in the morning. The amount of glycosilated polyphenols was assessed spectophotometrically at 280 nm, using synthetic catechin as standard. Glycosilated phloritzin, chlorogenic acid and quercetin were measured by HPCL-MS [high performance liquid chromatography-mass spectrometry].

The randomization was performed 1:1 ratio and the blocks were stratified by sex and age. An alphabetical code was assigned to each lot code (corresponding to treatment or placebo) impressed on the dose box. The study staffs and the investigators, as well as all of the volunteers, were blinded to the group assignment. Codes were kept in a sealed envelope, which was not opened until the end of the trial. Dose boxes were mixed and a blinded dose box was assigned to each enrolled patient.

Patients were evaluated anamnestically and by the execution of a physical examination and laboratory analyses at the baseline, in the middle and at the end of the trial.

The hemodynamic variables recorded (endothelial function, arterial stiffness and related parameters) were investigated before and after the intervention period. All the instrumental measurements were carried out following standardized protocols by specially trained staff.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI)>25 kg/m2
* Fasting plasma glucose 100 mg/dL ≤ FPG ≤ 125 mg/dL

Exclusion Criteria:

* Patients with obesity (body mass index [BMI] <30 Kg/m2)
* diabetes mellitus
* personal history of atherosclerosis-related cardiovascular diseases (coronary artery disease
* cerebrovascular disease
* ultrasound diagnosed carotid atherosclerosis)
* absorption disease
* myopathy
* renal failure or chronic liver disease
* serious or invalidating other diseases reducing the subjects' ability to comply with the full protocol were excluded from the study as well as subjects with a known apple intolerance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 8 week
  Change in arterial diameter after ischemic stimulus

CONTACTS AND LOCATIONS:
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cicero AFG, Caliceti C, Fogacci F, Giovannini M, Calabria D, Colletti A, Veronesi M, Roda A, Borghi C. Effect of apple polyphenols on vascular oxidative stress and endothelium function: a translational study. Mol Nutr Food Res. 2017 Nov;61(11). doi: 10.1002/mnfr.201700373. Epub 2017 Sep 1. PMID 28755406